CLINICAL TRIAL: NCT07277907
Title: Efficacy and Safety of Lubiprostone in the Treatment of Slow Transit Constipation: A Multicenter, Randomized Controlled Trial
Brief Title: Efficacy and Safety of Lubiprostone in the Treatment of Slow Transit Constipation
Acronym: STOPS 03
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Director, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LB20250919; 82370547 (Other Grant/Funding Number: National Natural Science Foundation of China Project)
Record Dates: First submitted 2025-09-28; First posted 2025-12-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Slow Transit Constipation; Pharmacotherapy
Keywords: Slow Transit Constipation; Lubiprostone; Polyethylene Glycol; Randomized Controlled Trial; medication
MeSH Terms: interventions — Lubiprostone; Polyethylene Glycols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lubiprostone (Experimental): Lubiprostone is an oral bicyclic fatty acid that selectively activates type 2 chloride channels in the apical membrane of human gastrointestinal epithelial cells, thereby increasing chloride-rich fluid secretion. Although the mechanism is unclear, this may then decrease intestinal transit time, allowing the passage of stool and alleviating symptoms of constipation.
  Interventions: Drug: Lubiprostone
- Polyethylene Glycol (Active Comparator): Polyethylene glycol (PEG ) is an established osmotic laxative, widely available worldwide for the treatment of functional constipation in adults and children.
  Interventions: Drug: Polyethylene glycol (PEG )

INTERVENTIONS:
Drug: Lubiprostone — Patients were instructed to orally ingest Lubiprostone Soft Capsules (provided by Nanjing Chia-Tai Tianqing Pharmaceutical Company) at a dose of 24 μg twice daily with food and water during breakfast and dinner. The capsules must be swallowed whole without splitting or chewing. The treatment duration was 4 weeks, and medication adherence was monitored through patient diaries and pill count of returned medication.
  Arms: Lubiprostone
Drug: Polyethylene glycol (PEG ) — Subjects in the control group will receive the standard treatment of polyethylene glycol 4000 powder at a dosage of 10 g, twice daily. Each dose will be dissolved in 200-250 mL of water and administered orally for 4 weeks.
  Arms: Polyethylene Glycol

SUMMARY:
Lubiprostone has established efficacy and a favorable safety profile in chronic constipation and irritable bowel syndrome with constipation (IBS-C). However, clinical data specifically supporting its use in slow-transit constipation (STC), a distinct subtype of chronic constipation, remains limited.

DETAILED DESCRIPTION:
Slow-transit constipation (STC) is a common subtype of chronic constipation, accounting for up to 30% of cases. Its clinical hallmarks include a diminished or absent urge to defecate and a significantly reduced stool frequency (spontaneous bowel movements <3 per week). The condition often follows a prolonged and progressively worsening course, characterized by straining, passage of hard stools, and associated symptoms such as abdominal pain and bloating. In severe cases, fecal impaction and consequent colonic obstruction may occur, substantially impairing the patient's quality of life.

Non-surgical management, including lifestyle modifications, pharmacological therapy, gut microbiome modulation, and sacral nerve stimulation, remains the first-line approach for most STC patients. Among these, pharmacotherapy is central. Conventional agents include bulk-forming, osmotic, and stimulant laxatives, as well as prokinetics. However, these options are often limited by adverse effects-such as abdominal pain, bloating, rash, drug dependence, malabsorption, and electrolyte imbalances-and the development of tolerance with long-term use. This frequently leaves patients with inadequate relief, creating an urgent need for more effective and safer therapeutics.

Lubiprostone, a chloride channel activator that functions as a secretagogue, enhances intestinal fluid secretion and motility. Its efficacy and safety in chronic idiopathic constipation and irritable bowel syndrome with constipation are well-documented, leading to approvals by the U.S. FDA for these indications. Nevertheless, specific data on its use for STC, a distinct pathophysiological entity, is lacking. This study is therefore designed to evaluate the clinical efficacy and safety of lubiprostone in an STC population, with the aim of generating new evidence to inform precise treatment strategies for this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in the study and provided signed informed consent;
2. Met the Rome IV diagnostic criteria for functional constipation;
3. Had fewer than 3 spontaneous bowel movements (SBMs) per week;
4. More than 20% the radio-paque markers localized in the colon after 72 hours based on colonic transit studies;
5. Were able to complete the bowel movement diary and study questionnaires as required by the study protocol;
6. Agreed to use effective contraception from the time of signing the informed consent form until 3 months after the last dose of the study drug;
7. Aged 18 years or older, both males and females.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with severe outlet obstruction constipation (e.g. Oxford Grade IV or above for rectal prolapse, rectocele > 3.1 cm, puborectalis syndrome).
3. Patients with hyperthyroidism or hypothyroidism.
4. Patients with opioid-induced constipation.
5. Patients with megacolon or megarectum.
6. Patients with apparent mechanical intestinal obstruction.
7. Patients with inflammatory bowel disease (e.g. Crohn's disease or ulcerative colitis).
8. Patients with malignant tumors of the digestive system.
9. Patients with a history of colorectal surgery.
10. Patients with a previous history of taking lubiprostone.
11. Patients with severe symptoms of depression or anxiety.
12. Patients with known or suspected hypersensitivity to lubiprostone/polyethylene glycol 4000 or any excipients.
13. Patients requiring medications for Parkinson's disease, antipsychotics, antimanic agents, or psychostimulants.
14. Patients with severe cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, neurological, or psychiatric diseases.
15. Other patients deemed by the investigator as unsuitable for participation in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The change in spontaneous bowel movements (SBMs) frequency from baseline during the first week | From 2 weeks prior to the first dose through 4 weeks after treatment initiation
  The change from baseline in the weekly average number of SBMs reported during the first week after treatment initiation

SECONDARY OUTCOMES:
The percentage of patients with SBMs within 24 hours after the first intake of the study drug | Day 1 after treatment initiation
Time to first SBM occurrence after treatment initiation | Up to 4 weeks after treatment initiation
The percentage of patients reporting 3 or more SBMs/wk | From 2 weeks prior to the first dose through 4 weeks after treatment initiation
The percentage of patients achieving an increase of ≥1 SBMs/week from baseline | From 2 weeks prior to the first dose through 4 weeks after treatment initiation
The change from baseline in the weekly average number of SBMs at weeks 2, 3, and 4 | From 2 weeks prior to the first dose through 4 weeks after treatment initiation
The change from baseline in the Bristol Stool Form Scale (BSFS) values for SBMs at weeks 1 and 4 | The 1 and 4-week treatment period has been completed
  The BSFS values can be described as the following 7 types: 1. separate hard lumps; 2. sausage-shaped but lumpy; 3. like a sausage but with cracks; 4. like a sausage, smooth and soft; 5. soft blobs with clear cut edges; 6. a mushy stool; and 7. watery.
The change from baseline in the ratings of straining associated with SBMs at weeks 1 and 4 | The 1 and 4-week treatment period has been completed
  The ratings of straining will be described using a 5-point Likert scale: 0= absent; 1= mild; 2= moderate; 3= severe; and 4= very severe
The change from baseline in the Wexner constipation score at weeks 1 and 4 | The 1 and 4-week treatment period has been completed
  The Wexner Constipation Score will be recorded in terms of scores. Questions examine constipation in its clinical expressions. Each question is answered on a scale of 0 to 4. The scale ranges from 0 (best) to 30 (worst)
The change from baseline in the Patient Assessment of Constipation Quality of Life (PAC-QOL) score at weeks 1 and 4 | The 1 and 4-week treatment period has been completed
  The full PAC-QOL consists of 28 items rated on a 5-point Likert scale ("1" = Not at all / None of the time; "2" = A little bit / A little of the time; "3" = Moderately /Some of the time; "4" = Quite a bit / Most of the time; "5" = Extremely / All of the time)
The patients' satisfaction scores at weeks 1 and 4 | The 1 and 4-week treatment period has been completed
  The patients' satisfaction scores will be described using a 5-point Likert scale: 0= Not at all; 1= A little bit; 2= Moderately; 3= Quite a bit; and 4= Extremely
The rate of adverse reactions, including nausea, diarrhea, and abdominal pain. | Up to 4 weeks after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Tong, MD, Study Director — Army Medical Center (Daping Hospital)
Locations (15):
- China (15):
  - Bishan Hospital of Chongqing, Bishan, Chongqing Municipality
  - the People's Hospital of HeChuan Chongqing, Hechuan, Chongqing Municipality
  - Shapingba Hospital, Chongqing University, Shapingba, Chongqing Municipality
  - The Chenjiaqiao Hospital of ShaPingba District of Chongqing, Shapingba, Chongqing Municipality
  - Army Medical Center (Daping Hospital), Yuzhong, Chongqing Municipality
  - Gansu Province Central Hospital, Lanzhou, Gansu
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - General Hospital of the Eastern Theater Cammand of the PLA, Nanjing, Jiangsu
  - Renji Hospital, Shanghai Jiaotong University, Pudong, Shanghai Municipality
  - Xijing Hospital, Xi’an, Shanxi
  - Chengdu Analrectal Hospital, Chengdu, Sichuan
  - The General Hospital of Western Theater Command, Chengdu, Sichuan
  - The Second People's Hospital of Yibin, Yibin, Sichuan
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cinca R, Chera D, Gruss HJ, Halphen M. Randomised clinical trial: macrogol/PEG 3350+electrolytes versus prucalopride in the treatment of chronic constipation -- a comparison in a controlled environment. Aliment Pharmacol Ther. 2013 May;37(9):876-86. doi: 10.1111/apt.12278. Epub 2013 Mar 11. PMID 23480216
- [Result] Chang L, Chey WD, Imdad A, Almario CV, Bharucha AE, Diem S, Greer KB, Hanson B, Harris LA, Ko C, Murad MH, Patel A, Shah ED, Lembo AJ, Sultan S. American Gastroenterological Association-American College of Gastroenterology Clinical Practice Guideline: Pharmacological Management of Chronic Idiopathic Constipation. Gastroenterology. 2023 Jun;164(7):1086-1106. doi: 10.1053/j.gastro.2023.03.214. PMID 37211380
- [Result] Christie J, Shroff S, Shahnavaz N, Carter LA, Harrison MS, Dietz-Lindo KA, Hanfelt J, Srinivasan S. A Randomized, Double-Blind, Placebo-Controlled Trial to Examine the Effectiveness of Lubiprostone on Constipation Symptoms and Colon Transit Time in Diabetic Patients. Am J Gastroenterol. 2017 Feb;112(2):356-364. doi: 10.1038/ajg.2016.531. Epub 2016 Dec 6. PMID 27922028
- [Result] Li F, Fu T, Tong WD, Liu BH, Li CX, Gao Y, Wu JS, Wang XF, Zhang AP. Lubiprostone Is Effective in the Treatment of Chronic Idiopathic Constipation and Irritable Bowel Syndrome: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Mayo Clin Proc. 2016 Apr;91(4):456-68. doi: 10.1016/j.mayocp.2016.01.015. PMID 27046523
- [Result] Jamal MM, Adams AB, Jansen JP, Webster LR. A randomized, placebo-controlled trial of lubiprostone for opioid-induced constipation in chronic noncancer pain. Am J Gastroenterol. 2015 May;110(5):725-32. doi: 10.1038/ajg.2015.106. Epub 2015 Apr 28. PMID 25916220
- [Result] Ondo WG, Kenney C, Sullivan K, Davidson A, Hunter C, Jahan I, McCombs A, Miller A, Zesiewicz TA. Placebo-controlled trial of lubiprostone for constipation associated with Parkinson disease. Neurology. 2012 May 22;78(21):1650-4. doi: 10.1212/WNL.0b013e3182574f28. Epub 2012 May 9. PMID 22573627
- [Result] Chey WD, Drossman DA, Johanson JF, Scott C, Panas RM, Ueno R. Safety and patient outcomes with lubiprostone for up to 52 weeks in patients with irritable bowel syndrome with constipation. Aliment Pharmacol Ther. 2012 Mar;35(5):587-99. doi: 10.1111/j.1365-2036.2011.04983.x. Epub 2012 Jan 18. PMID 22251419
- [Result] Carter NJ, Scott LJ. Lubiprostone: in constipation-predominant irritable bowel syndrome. Drugs. 2009 Jun 18;69(9):1229-37. doi: 10.2165/00003495-200969090-00007. PMID 19537839
- [Result] Fukudo S, Hongo M, Kaneko H, Takano M, Ueno R. Lubiprostone increases spontaneous bowel movement frequency and quality of life in patients with chronic idiopathic constipation. Clin Gastroenterol Hepatol. 2015 Feb;13(2):294-301.e5. doi: 10.1016/j.cgh.2014.08.026. Epub 2014 Aug 24. PMID 25158925
- [Result] Cryer B, Katz S, Vallejo R, Popescu A, Ueno R. A randomized study of lubiprostone for opioid-induced constipation in patients with chronic noncancer pain. Pain Med. 2014 Nov;15(11):1825-34. doi: 10.1111/pme.12437. Epub 2014 Apr 9. PMID 24716835
- [Result] Lang L. The Food and Drug Administration approves lubiprostone for irritable bowel syndrome with constipation. Gastroenterology. 2008 Jul;135(1):7. doi: 10.1053/j.gastro.2008.06.004. Epub 2008 Jun 9. No abstract available. PMID 18541153
- [Result] Johanson JF, Morton D, Geenen J, Ueno R. Multicenter, 4-week, double-blind, randomized, placebo-controlled trial of lubiprostone, a locally-acting type-2 chloride channel activator, in patients with chronic constipation. Am J Gastroenterol. 2008 Jan;103(1):170-7. doi: 10.1111/j.1572-0241.2007.01524.x. Epub 2007 Oct 4. PMID 17916109
- [Result] Sweetser S, Busciglio IA, Camilleri M, Bharucha AE, Szarka LA, Papathanasopoulos A, Burton DD, Eckert DJ, Zinsmeister AR. Effect of a chloride channel activator, lubiprostone, on colonic sensory and motor functions in healthy subjects. Am J Physiol Gastrointest Liver Physiol. 2009 Feb;296(2):G295-301. doi: 10.1152/ajpgi.90558.2008. Epub 2008 Nov 25. PMID 19033530
- [Result] Crowell MD. Lubiprostone: trials and tribulations. Nat Rev Gastroenterol Hepatol. 2009 May;6(5):259-60. doi: 10.1038/nrgastro.2009.62. No abstract available. PMID 19404263
- [Result] Sajid MS, Hebbar M, Baig MK, Li A, Philipose Z. Use of Prucalopride for Chronic Constipation: A Systematic Review and Meta-analysis of Published Randomized, Controlled Trials. J Neurogastroenterol Motil. 2016 Jul 30;22(3):412-22. doi: 10.5056/jnm16004. PMID 27127190
- [Result] Lee-Robichaud H, Thomas K, Morgan J, Nelson RL. Lactulose versus Polyethylene Glycol for Chronic Constipation. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007570. doi: 10.1002/14651858.CD007570.pub2. PMID 20614462
- [Result] Vlismas LJ, Wu W, Ho V. Idiopathic Slow Transit Constipation: Pathophysiology, Diagnosis, and Management. Medicina (Kaunas). 2024 Jan 6;60(1):108. doi: 10.3390/medicina60010108. PMID 38256369
- [Result] Mohaghegh Shalmani H, Soori H, Khoshkrood Mansoori B, Vahedi M, Moghimi-Dehkordi B, Pourhoseingholi MA, Norouzinia M, Zali MR. Direct and indirect medical costs of functional constipation: a population-based study. Int J Colorectal Dis. 2011 Apr;26(4):515-22. doi: 10.1007/s00384-010-1077-4. Epub 2010 Oct 19. PMID 20957375
- [Result] Rao SS, Rattanakovit K, Patcharatrakul T. Diagnosis and management of chronic constipation in adults. Nat Rev Gastroenterol Hepatol. 2016 May;13(5):295-305. doi: 10.1038/nrgastro.2016.53. Epub 2016 Apr 1. PMID 27033126
- [Result] Bharucha AE, Pemberton JH, Locke GR 3rd. American Gastroenterological Association technical review on constipation. Gastroenterology. 2013 Jan;144(1):218-38. doi: 10.1053/j.gastro.2012.10.028. No abstract available. PMID 23261065
- [Result] Bharucha AE, Lacy BE. Mechanisms, Evaluation, and Management of Chronic Constipation. Gastroenterology. 2020 Apr;158(5):1232-1249.e3. doi: 10.1053/j.gastro.2019.12.034. Epub 2020 Jan 13. PMID 31945360